CLINICAL TRIAL: NCT06856369
Title: Clinical Efficacy of 1% Metformin and Alendronate Gel in Adjunct to Fibrin in Chronic Periodontitis
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Bahria University (Other)
Collaborators: Islamabad Medical and Dental College (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BUHS-IRB#125/24
Record Dates: First submitted 2025-02-10; First posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-01

CONDITIONS: Alveolar Bone Loss Associated Chronic Periodontitis
Keywords: chronic periodontitis; intra-bony defect depth; metformin; alendronate; platelet rich fibrin
MeSH Terms: conditions — Chronic Periodontitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Platelet Rich Fibrin (Active Comparator): Group A - administration of Platelet rich fibrin only, subgingivally , once in 6 months
  Interventions: Procedure: Platelet rich fibrin
- Metformin (Active Comparator): Group -B - Platelet Rich Fibrin +1% Metformin gel, once sub-gingivally in 6 months
  Interventions: Drug: Metformin hydrochloride powder
- Alendronate (Active Comparator): Group C- Platelet rich fibrin + 1% Alendronate gel , once sub-gingivally in 6 months
  Interventions: Drug: alendronate sodium powder

INTERVENTIONS:
Procedure: Platelet rich fibrin — sub-gingival administration of platelet rich fibrin following open flap surgery
  Arms: Platelet Rich Fibrin
Drug: Metformin hydrochloride powder — subgingival administration of 1% Metformin Hydrochloride gel with platelet rich fibrin following open flap surgery
  Arms: Metformin
Drug: alendronate sodium powder — subgingival administration of 1% Alendronate gel with platelet rich fibrin following open flap surgery
  Arms: Alendronate

SUMMARY:
This open label, randomized controlled clinical trial study will be conducted after obtaining ERC approval of Bahria University Health Sciences. Written informed consent will be taken from all study participants. Patients suffering from moderate to severe chronic periodontitis and diagnosed as per criteria Community Periodontal Index for Treatment Needs (CPITN) (Heiko Z et al, 2015) will be selected from the Oral Diagnostic & Periodontology department of Islamabad Medical & Dental College hospital . Patients will be randomized into 3 groups by using computer driven list. Sample size will be calculated by using software G power version3.1.9.2 . Patients will be randomly divided into 3 groups.

(I) Baseline investigations/parameters (at day zero): FBS values will be monitored using digital glucometer Clinical parameters (PI, CAL, PDD, mSBI) will be assessed at baseline, 3 , 6 , 9 & 12 months by calibrated periodontal probe. Radiological parameters (VBL & IBDA) will be carried out using OPG at baseline, 6 & 12 months. ELISA for Transforming growth factor (TGFβ) and osteocalcin biomarkers will be done at baseline and 3 months. RT-PCR for the detection of RUNX2 gene will be done at baseline and 3 months Patient will be called at 14th day for suture removal and clinical assessment . Follow up will be done at 3, 6, 9 and 12 months to assess clinically. Radiographic parameters will be assessed at 6 &12 months. Pharmacogenetic parameters will be assessed at 6months. All patients will be advised regular check-ups post surgically at per appointment . Individual study period will be 12 months. Total duration of study will be 15 months.

Primary outcomes:

Reduction in intra-bony defect angle and vertical bone loss. Periodontal and alveolar bone regeneration by detecting the levels of biomarkers namely, transforming growth factor β, osteocalcin

Secondary Outcomes:

Osteogenic proliferation : Evaluation of RUNX2 expression in response to Metformin & Alendronate 1% gel administration will be assessed per subject per genetic analysis.

RUNX2 expression will be observed through RT- PCR.

DETAILED DESCRIPTION:
This open -label randomized controlled clinical trial study will be conducted after obtaining IRB approval of Bahria University Health Sciences Campus, Karachi. Written informed consent will be taken from all study participants. Patients suffering from moderate to severe chronic periodontitis and diagnosed as per criteria Community Periodontal Index for Treatment Needs (CPITN) will be selected from the Oral Diagnostic & Periodontology department of Islamabad Medical & Dental College. Patients will be randomized into 3 groups by using computer driven list.

A. Group A: PRF alone (Control group, n=40) B. Group B: 1% Metformin gel + PRF (test group,n=40) C. Group C : 1% Alendronate gel + PRF (test group,n=40) Clinical examination will be done at baseline, 3,6,9 & 12 months by means of periodontal probe assessing PDD, CAL, mSBI, PI for the diagnosis of chronic periodontitis. Radiological parameters ( VBL, IBDDR & IBDA) will be carried out using orthopantamogram at baseline and 6 months. Patients will be advised not to eat 2 hours prior treatment . Paper points #30 (GAPADENT) sterilized colour coded will be used for the collection of gingival crevicular fluid from the crevicular site. Selected affected tooth with deep periodontal pocket and clinical attachment loss will be isolated with cotton rolls to prevent salivary contamination, supra-gingival plaque will be removed without disturbing the soft tissues, and the tooth will be dried with a gentle stream of air for 5s. Gingival crevicular fluid will preferably be collected by absorption technique from the affected tooth. Absorbent paper points #30 will be standardized to three in quantity for Gingival crevicular fluid sampling. These will be placed into the periodontal pocket of the affected tooth with the greatest pocket depth (≥4mm) in each patient till mild resistance is felt. The paper points were left for 30 seconds to collect the resting GCF. The paper points contaminated with blood or saliva will be discarded .The sample will be transferred to Eppendorf tubes (2 ml) containing 150 µl phosphate-buffered saline (PBS; Sigma Aldrich, St. Louis, M) , centrifuged at 10,000 Rev/min for 5 mins and stored at -800C 14. Genotyping- DNA sequence variation for RUNX2 will be done by real time PCR.14, 25. Transforming growth factor-β (TGF-β) and osteocalcin will be assessed by ELISA. Intra- sulcular incision with mucoperiosteal flap elevation, debridement of granulation tissue, subgingival SRP, and rinsing with normal saline solution will be performed. For the prepaartion of PRF Intravenous blood from the antecubital vein will be collected in three, 10-ml sterilized test tubes. No anticoagulant will be added to the tubes and instantly centrifuged in centrifugation machine at 3000 RPM for 10 min. The formation of structured fibrin clot in the centre of the tube, just in the middle of the red corpuscles at the base and acellular plasma (platelet-poor plasma [PPP]) at the top. PRF will be separated from RBCs using sterile tweezers and scissors just after the removal of PPP. Then, it will be transferred onto sterile gauze , compress so as to squeeze out the serum out of a stable PRF membrane. This membrane will be placed at the site along with gel administration by means of syringe. Group A (control) will undergo open flap debridement (OFD) with platelet rich fibrin (PRF) only, Group B will have OFD with administration of 1% Metformin gel in adjunct to PRF and Group C will have OFD with administration of 1% Alendronate gel in adjunct to PRF. Patient will be called for suture removal at day 14. Follow up will be done at 3, 6, 9 & 12 months to assess clinical parameters . Biochemical and pharmacogenetic parameters will be assessed 3 months . Radiographic parameters will be assessed at 6 & 9 months. All patients will be advised regular check-ups post surgically . Data analysis will be performed by statistical software package SPSS version 23. The frequencies and percentages will be calculated for categorical data while mean with standard deviation will be calculated for continuous characteristics. Intra-group comparison will be analysed by paired Student's t-test. Inter-group comparison analysis will be done by ANOVA. Multiple comparison analysis will be performed by Post Hoc. P-value < 0.05 is considered significant.

ELIGIBILITY:
Inclusion Criteria:

* • Males and females

  * Age 25-50 years
  * Systemically healthy individuals
  * Probing depth sites ≥ 5mm- <7 mm pocket depth (PD)[American Dental Association/ Academy of Periodontology 1999) Clinical attachment level (CAL) ≥4mm- <5 mm [ American Dental Association/ Academy of Periodontology 1999)
  * Vertical bone loss (VBL) ≥3mm on intraoral periapical radiographs.[American Academy of Periodontology Guidelines, 1999]
  * Modified Sulcus bleeding index (mSBI) [Muhlemann and Sons index,1971; Augusta B Rebelo et al,2011]
  * No history of periodontal treatment in the previous 6 months

Exclusion Criteria:

* • Individuals <20 and >50 yrs

  * Patients with known systemic disease such as diabetes, hypertension, osteoporosis etc.
  * Patients with severe periodontitis
  * Pregnant and lactating mothers
  * Patients receiving medications

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2025-01-22 (Actual); Primary Completion 2026-02-14 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Reduction in intra-bony defect depth in millimeters in patients suffering from chronic periodontitis | 6, 9 & 12 months
  Assessment will be done at 6, 9 & 12 months using Orthopantomogram

SECONDARY OUTCOMES:
Osteogenic proliferation | 3 months
  Evaluation of RUNX2 expression in response to Metformin & Alendronate 1% gel administration will be assessed per subject per genetic analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Mamoora Arslaan, MPhil, Principal Investigator — Bahria University Islamabad
Locations (1):
- Islamabad Medical & Dental College, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
All data will be shared
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The IPD data will become accessible one year after publication and will remain available indefinitely
Access Criteria: all data will be accessible to every one

REFERENCES:
- [Result] Arena C, Caponio VCA, Zhurakivska K, Lo Russo L, Lo Muzio L, Troiano G. Added effect of 1% topical alendronate in intra-bony and inter-radicular defects as part of step II periodontal therapy: a systematic review with meta-analysis and trial sequential analysis. BMC Oral Health. 2022 Jan 21;22(1):15. doi: 10.1186/s12903-022-02044-1. PMID 35062940
- [Result] Ozcan E, Saygun I, Kantarci A, Ozarslanturk S, Serdar MA, Ozgurtas T. The effects of a novel non-invasive application of platelet-rich fibrin on periodontal clinical parameters and gingival crevicular fluid transforming growth factor-beta and collagen-1 levels: A randomized, controlled, clinical study. J Periodontol. 2021 Sep;92(9):1252-1261. doi: 10.1002/JPER.20-0713. Epub 2021 Jan 15. PMID 33382101
- [Result] Hu J, Han J, Jin M, Jin J, Zhu J. Effects of metformin on bone mineral density and bone turnover markers: a systematic review and meta-analysis. BMJ Open. 2023 Jun 23;13(6):e072904. doi: 10.1136/bmjopen-2023-072904. PMID 37355276
- [Result] Chang J, Blanchard SB, Windsor LJ, Gregory RL, Hamada Y. Levels of growth factors from platelet-rich fibrin from chronic periodontitis versus periodontally healthy subjects: a pilot study. Clin Oral Investig. 2020 Feb;24(2):823-832. doi: 10.1007/s00784-019-02944-7. Epub 2019 Jun 13. PMID 31197657
- See also: PMID: 35062940 — https://pubmed.ncbi.nlm.nih.gov/35062940/